CLINICAL TRIAL: NCT01285726
Title: Initiative for Patient Outcomes in Dialysis - PD (IPOD-PD Study)
Brief Title: Initiative for Patient Outcomes in Dialysis - Peritoneal Dialysis (PD) (IPOD-PD Study)
Acronym: IPOD-PD
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: BCM-PD-02-INT
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Renal Failure
Keywords: Peritoneal dialysis; Hydration status; Residual renal function; Bioimpedance spectroscopy; Body composition monitor
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non-interventional study — This is a purely non-interventional, observational study, where treatment decisions are completely guided by the discretion of the attending nephrologists.

SUMMARY:
The aim of the study is to asses the hydration status of incident peritoneal dialysis (PD) patients and its evolution over a period of four years, independent of the PD treatment modality (APD or CAPD) and the PD solution type.

DETAILED DESCRIPTION:
Achieving optimal fluid balance remains a major clinical challenge in peritoneal dialysis (PD) patients. With the recent development of a new bioimpedance spectroscopy (BIS) device, the BCM-Body Composition Monitor (BCM), it is now possible to quantify deviations of hydration status and to define target weight directly.

It has been observed that more than 50% of the PD patients are overhydrated, as compared to the healthy population. This overhydration seems to be associated with modifiable practice-related factors, such as correct PD prescription according to membrane transport status, and dietary fluid intake.

The aim of this study is to assess the hydration status of incident PD patients, and diagnose the underlying reasons for incorrect fluid status. In addition, changes in fluid status, residual renal function and nutritional status, over a follow-up period of up to four years will be registered.

The investigators assume that the use of the BCM-Body Composition Monitor (BCM) provides quantitative measurement of hydration status and thereby supports physicians in identifying patients who are not euvolaemic. Hence, the BCM allows an improved management of underlying causes of non-euvolaemic hydration state and appropriate monitoring of fluid status.

ELIGIBILITY:
Inclusion Criteria:

* Incident patients directly before start of peritoneal dialysis
* Patients in whom routine measurement of body composition monitoring is performed

Exclusion Criteria:

* Patients treated with HD before start of PD
* Patients in whom body composition monitoring cannot be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic kidney disease (CKD) starting renal replacement therapy on APD or CAPD
Sampling Method: Non-Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hydration status | Every three months over a period of four years
  Assessed via body composition measurements (Overhydration, total body water (TBW), extracellular water (ECW), intracellular water (ICW)) (Overhydration, total body water (TBW), extracellular water (ECW), intracellular water (ICW))

SECONDARY OUTCOMES:
Residual renal function | Every three months over a period of four years
Peritoneal transport status | Every three months over a period of four years
Time to change to haemodialysis | Four years
Changes in PD prescription | Four years

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, Prof, Study Chair — Ospedale San Bartolo; Wim Van Biesen, Prof, Study Chair — University Hospital, Ghent; Christian Verger, Dr, Study Chair — French Language PD Registry (RDPLF)
Locations (134):
- Klinikum Wels, Wels, Austria
- Belgium (6):
  - ASZ Aalst, Aalst
  - ASZ Geraardsbergen, Geraardsbergen
  - Ghent University Hospital, Ghent
  - U.Z. Leuven, Leuven
  - CHU Sart Tilman, Liège
  - Heilig-Hart Roeselare, Roeselare
- Bosnia and Herzegovina (2):
  - KBC Mostar, Mostar
  - UKC Tuzla, Tuzla
- Brazil (3):
  - Instituto Mineiro Nefrologia, Belo Horizonte
  - CDR Barra do Piraí, Piraí
  - CETENE, São Paulo
- Croatia (3):
  - UHC Osijek, Osijek
  - UH Split, Split
  - UH Merkur, Zagreb
- Instituto de Nefrología, La Habana, Cuba
- Czechia (7):
  - University Hospital FN Brno Bohunice, Brno
  - FN Hradec Kralove, Hradec Králové
  - DS Most, Most
  - Faculty Hospital Plzen, Pilsen
  - IKEM, Prague
  - VFN Strahov, Prague
  - Třebíč Hospital, Třebíč
- Denmark (3):
  - Herlev Hospital, Herlev
  - Hillerød Hospital, Hillerød
  - Roskilde Hospital, Roskilde
- Estonia (3):
  - North Estonian Regional Hospital, Tallinn
  - West Talinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Finland (7):
  - Helsinki University Hospital, Helsinki
  - Central Hospital in Joensuu, Joensuu
  - Keski-Suomen keskussairaala, Jyväskylä, Jyväskylä
  - Kymenlaakson keskussairaala, Kotka, Kotka
  - Oulu University Hospital, Oys
  - Satakunnan keskussairaala, Pori, Pori
  - Tampere University Hospital, Tampere
- France (7):
  - CHU de Bordeaux, Bordeaux
  - C.H. Dunkerque, Dunkirk
  - Hôpital Bichat - Claude Bernard, Paris
  - Centre Hospitalier René Dubos, Pontoise
  - AUB Quimper / Centre Hospitalier Laennec, Quimper
  - ECHO Confluent, Rezé
  - Hôpital Civil de Strasbourg, Strasbourg
- Germany (7):
  - KfH Nierenzentrum Bottrop, Bottrop
  - Klinikum Braunschweig, Braunschweig
  - Nierenzentrum Heidelberg, Heidelberg
  - Nieren und Hochdruckzentrum Kiel, Kiel
  - Robert Bosch Krankenhaus, Stuttgart
  - Nephrologisches Zentrum Velbert Innere Medizin und Nephrologie, Velbert
  - Nephrologische Praxis Wiesbaden, Wiesbaden
- Greece (5):
  - General University Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens G. Gennimatas, Athens
  - General Hospital of Ioannina, Ioannina
  - General University Hospital of Ioannina, Ioannina
  - General University Hospital of Thessaloniki "AHEPA", Thessaloniki
- MMM - Chennai, Chennai, India
- Western Galilee Hospital, Nahariya, Israel
- Italy (4):
  - UO Nefrologia Policlinico BARI, Bari
  - Azienda Ospedaliera Brotzu, Cagliari
  - Ospedale Civico Palermo, Palermo
  - Ospedale San Bartolo, Vicenza
- Latvia (2):
  - Med Alfa Ltda, Riga
  - P. Stradins hospital, Riga
- Lithuania (3):
  - Kaunas clinics, Kaunas
  - Klaipeda Republic Hospital, Klaipėda
  - Vilnius Univ. Antakalnio Hospital, Vilnius
- University Hospital Maastricht, Maastricht, Netherlands
- Norway (4):
  - Sykehuset i Møre og Romsdal HF, Ålesund
  - Nordlandssykehuset Bodø, Bodø
  - Sykehuset Levanger, Levanger
  - St. Olavs Hospital, Sluppen
- Portugal (2):
  - Hospital Santa Cruz, Carnaxide
  - CHP Hospital Santo Antonio, Porto
- South Korea (5):
  - Yeungnam University Hospital, Daegu
  - NHIC Ilsan Hospital, Goyang
  - Konkuk University Medical Center, Seoul
  - Seoul National University Hospitall, Seoul
  - Severance Hospital, Seoul
- Spain (34):
  - Hospital Universitario A Coruñ, A Coruña
  - CHU Albacete, Albacete
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hospital De Torrecardenas, Almería
  - Fundació Puigvert, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital de Galdakano, Bilbao
  - Hospital Univ. Puerta del Mar, Cadiz
  - Hospital General de Castellón, Castellon
  - Hospital Josep Trueta, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - CAULE, León
  - Hospital San Pedro, Logroño
  - Hospital Lucus Augusti, Lugo
  - Fundación Jiménez Díaz, Madrid
  - HGU Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Severo Ochoa, Madrid
  - Hospital Univ. Ramón y Cajal, Madrid
  - Hospital Universitario Puerta, Madrid
  - Fundación Hospital Manacor, Manacor
  - Hospital Carlos Haya, Málaga
  - Hospital de Mollet, Mollet del Vallès
  - Hospital Universitario Central, Oviedo
  - Hospital Univ. de Puerto Real, Puerto Real
  - HUM Valdecilla, Santander
  - CHUS, Santiago de Compostela
  - Hospital Virgen de la Macarena, Seville
  - Hospital Clínico de Valencia, Valencia
  - Hospital Rio Hortega, Valladolid
  - Hospital general de Vic, Vic
  - CHU Xeral Cies Vigo, Vigo
  - Hospital Txagorritxu, Vitoria-Gasteiz
- Sweden (8):
  - Mälarsjukhuset Eskilstuna, Eskilstuna
  - Sahlgrenska PD-mottagningen, Gothenburg
  - Hallands Hospital Halmstad, Halmstad
  - Sunderby Sjukhus, Luleå
  - Skånes Universitetssjukhus Malmo, Malmo
  - Danderyds Hospital, Stockholm
  - Karolinska Univers. Hospital, Stockholm
  - Kungsholmsdialysen, Stockholm
- Luzern Kantonsspital, Lucerne, Switzerland
- Akdeniz Universitesi, Antalya, Turkey (Türkiye)
- United Kingdom (2):
  - Western Infirmary Glasgow, Glasgow
  - Royal London Hospital, London
- Venezuela (10):
  - FME Caracas, Caracas
  - FME Charallave, Charallave
  - Cenesuca (FME Cumana), Cumaná
  - FMC El tigre Edo Anzoátegui, El Tigre
  - FME Zulia, Maracaibo
  - FME Maturin, Maturín
  - FME Puerto de la Cruz, Puerto Cruz
  - FME Maracay, Turmero
  - Instituto Docente de Urologia, Valencia
  - Nefrologico Valencia sur, Valencia

REFERENCES:
- [Derived] Verger C, Ronco C, Van Biesen W, Heaf J, Vrtovsnik F, Vera Rivera M, Puide I, Azar R, Gauly A, Atiye S, De Los Rios T. Association of Prescription With Body Composition and Patient Outcomes in Incident Peritoneal Dialysis Patients. Front Med (Lausanne). 2021 Dec 24;8:737165. doi: 10.3389/fmed.2021.737165. eCollection 2021. PMID 35004718
- [Derived] Ronco C, Verger C, Crepaldi C, Pham J, De Los Rios T, Gauly A, Wabel P, Van Biesen W; IPOD-PD Study Group. Baseline hydration status in incident peritoneal dialysis patients: the initiative of patient outcomes in dialysis (IPOD-PD study)dagger. Nephrol Dial Transplant. 2015 May;30(5):849-58. doi: 10.1093/ndt/gfv013. Epub 2015 Mar 11. PMID 25762355